CLINICAL TRIAL: NCT03370913
Title: A Phase 3 Open-Label, Single-Arm Study To Evaluate The Efficacy and Safety of BMN 270, an Adeno-Associated Virus Vector-Mediated Gene Transfer of Human Factor VIII in Hemophilia A Patients With Residual FVIII Levels ≤ 1 IU/dL Receiving Prophylactic FVIII Infusions
Brief Title: Single-Arm Study To Evaluate The Efficacy and Safety of Valoctocogene Roxaparvovec in Hemophilia A Patients (BMN 270-301)
Acronym: BMN 270-301
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 270-301; 2017-003215-19 (EudraCT Number)
Record Dates: First submitted 2017-11-27; First posted 2017-12-13 (Actual); Results first posted 2023-11-28 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Hemophilia A
Keywords: Gene Therapy; Clotting Disorders; Blood Disorder; Blood Coagulation Disorders; Inherited Blood Coagulation disorders; Hematologic Diseases; Coagulation Protein Disorders; Hemorrhagic Disorders; Genetic Diseases; Inborn; Factor VIII; Coagulants
MeSH Terms: conditions — Hemophilia A; Hemostatic Disorders; Hematologic Diseases; Blood Coagulation Disorders; Blood Coagulation Disorders, Inherited; Coagulation Protein Disorders; Hemorrhagic Disorders; Genetic Diseases, Inborn | interventions — Valoctocogene Roxaparvovec

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- valoctocogene roxaparvovec Open Label (Experimental): Single administration of valoctocogene roxaparvovec at a dose of 6E13 vg/kg
  Interventions: Biological: valoctocogene roxaparvovec

INTERVENTIONS:
Biological: valoctocogene roxaparvovec — Adeno-Associated Virus Vector-Mediated Gene Transfer of Human Factor VIII in Hemophilia A
  Other Names: BMN 270

SUMMARY:
This Phase III clinical study will assess the impact of BMN 270 (compared to FVIII prophylaxis) on the number of bleeding episodes irrespective of exogenous FVIII replacement treatment in the efficacy evaluation period (EEP) (from Week 5 post-BMN 270 infusion (Study Day 33) or the end of FVIII prophylaxis plus the washout period (3 days for products of standard half-life or plasma-derived and 5 days for products of extended half-life), whichever is later, to last visit by the data cut-off for the 2-year analysis, hereafter referred to as "Post FVIII Prophylaxis to Last Visit"). The study will also assess the impact of BMN 270 (compared to FVIII prophylaxis) on: the number of bleeding episodes requiring exogenous FVIII treatment in "Post FVIII Prophylaxis to Last Visit", FVIII activity as measured by chromogenic sustrate assay at Week 104 following intravenous infusion of BMN 270, usage of exogenous FVIII replacement therapy in "Post FVIII Prophylaxis to Last Visit", health-related quality of life patient-reported outcomes at week 104 following intravenous infusion of BMN 270. The study will also evaluate the safety of the BMN 270.

ELIGIBILITY:
Inclusion Criteria:

1. Males ≥ 18 years of age with hemophilia A and residual FVIII levels ≤ 1 IU/dL as evidenced by medical history, at the time of signing the informed consent.
2. Must have been on prophylactic FVIII replacement therapy for at least 12 months prior to study entry.
3. Treated/exposed to FVIII concentrates or cryoprecipitate for a minimum of 150 exposure days (EDs).
4. No previous documented history of a detectable FVIII inhibitor, and results from a Bethesda assay or Bethesda assay with Nijmegen modification of less than 0.6 Bethesda Units (BU) on 2 consecutive occasions at least one week apart within the past 12 months.

Exclusion Criteria:

1. Detectable pre-existing antibodies to the adeno-associated virus 5 (AAV5) capsid.
2. Any evidence of active infection or any immunosuppressive disorder, except for HIV infection
3. Any evidence of active infection or any immunosuppressive disorder, including HIV infection (effective as of Protocol Amendment 3)
4. Significant liver dysfunction.
5. Prior liver biopsy showing significant fibrosis.
6. Evidence of any bleeding disorder not related to hemophilia A.
7. Platelet count of < 100 x 10^9/L.
8. Creatinine ≥ 1.5 mg/dL.
9. Liver cirrhosis of any etiology as assessed by liver ultrasound.
10. Chronic or active hepatitis B.
11. Active Hepatitis C.
12. Active malignancy, except non-melanoma skin cancer.
13. History of hepatic malignancy.
14. History of arterial or venous thromboembolic events.
15. Known inherited or acquired thrombophilia, including conditions associated with increased thromboembolic risk, such as atrial fibrillation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Biological males only
Enrollment: 144 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2020-11-16 (Actual); Study Completion 2024-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — BioMarin Pharmaceutical
Locations (49):
- United States (15):
  - Los Angeles Orthopedic Hospital, Orthopedic Hemophilia Treatment Center, Los Angeles, California
  - UC Davis Hemophilia Treatment Center, Sacramento, California
  - University of California San Diego, Hematology and Oncology, Hemophilia &Thrombosis Treatment Center, San Diego, California
  - UCSF Medical Center, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - St. Joseph's Children's Hospital, Center for Bleeding and Clotting Disorders, Tampa, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Department of Hematology, Chicago, Illinois
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Tulane University Hematology & Medical Oncology, New Orleans, Louisiana
  - University of Michigan, Pediatric Hematology and Oncology, Ann Arbor, Michigan
  - Wayne State University, Detroit Medical Center, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine, Department of Pediatrics, Division of Hematology/Oncology, St Louis, Missouri
  - UNC Hemophilia and Thrombosis Center, Chapel Hill, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
- Australia (5):
  - The Royal Adelaide Hospital (RAH), Adelaide
  - Royal Brisbane and Women's Hospital, Brisbane
  - Alfred Hospital, Melbourne
  - Fiona Stanley Hospital, Perth
  - Royal Prince Alfred Hospital, Sydney
- University Hospital Leuven, Leuven, Belgium
- Brazil (5):
  - Campinas Estadual University (UNICAMP) / Campinas Hemocentro / Hematologia E Hemoterapia Center, Campinas
  - Parana's Hematology And Hemotherapy Center (HEMEPAR), Curitiba
  - Arthur De Siqueira Cavalcanti Hematology State Institute, Rio de Janeiro
  - Sao Paulo University Clinical Hospital, São Paulo
  - Holy Spirit Hematology and Hemotherapy Center, Vitória
- France (2):
  - Regional University Hospital of Lille (CHRU de Lille), Lille
  - Hopital de la Timone Marseille - Assistance Publique des Hopitaux de Marseille, Marseille
- Germany (2):
  - Vivantes Clinic im Friedrichshain- Landsberger Allee, Berlin
  - University Clinic Bonn, Bonn
- Chaim Sheba Medical Center, Ramat Gan, Israel
- Maggiore Polyclinic Hospital, IRCCS Ca' Granda, Center for Hemophilia and Thrombosis Angelo Bianchi Bonomi, Milan, Italy
- Charlotte Maxeke Johannesburg Academic Hospital, Hemophilia Comprehensive Care Center, Johannesburg, South Africa
- Department of Pediatrics, Kyung Hee University Hospital at Gangdong, Seoul, South Korea
- Spain (2):
  - Hospital Teresa Herrera, A Coruña
  - University Hospital Virgen del Rocio (HUVR), Seville
- Taiwan (5):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Tri-Service General Hospital, Taipei
- United Kingdom (8):
  - Queen Elizabeth Hospital, Birmingham
  - Addenbrookes Hospital, Cambridge
  - Glasgow Royal Infirmary, Department of Hematology, Glasgow
  - Barts and The London School of Medicine and Dentistry, Haemophilia Centre, London
  - Hammersmith, London
  - St Thomas' Hospital, London
  - Churchill Hospital, Oxford Hemophilia and Thrombosis Center, Oxford
  - University Hospital Southampton NHS Foundation Trust, Southampton

REFERENCES:
- [Derived] Santos S, Robinson TM, Trueman D. Estimated Long-Term Durability of Valoctocogene Roxaparvovec Treatment in Male patients with Severe Hemophilia A: An Extrapolation of Clinical Data. Adv Ther. 2025 Nov;42(11):5781-5793. doi: 10.1007/s12325-025-03368-4. Epub 2025 Sep 23. PMID 40986187
- [Derived] Agarwal S, Sandza K, Obrochta Moss K, Vora M, Bowen A, Bunch B, Holcomb J, Robinson TM, Jayaram K, Russell CB, Zoog S, Vettermann C, Henshaw J. Blood biodistribution and vector shedding of valoctocogene roxaparvovec in people with severe hemophilia A. Blood Adv. 2024 Sep 10;8(17):4606-4615. doi: 10.1182/bloodadvances.2024013150. PMID 39024543
- [Derived] Oldenburg J, Chambost H, Liu H, Hawes C, You X, Yang X, Newman V, Robinson TM, Hatswell AJ, Hinds D, Santos S, Ozelo M. Comparative Effectiveness of Valoctocogene Roxaparvovec and Prophylactic Factor VIII Replacement in Severe Hemophilia A. Adv Ther. 2024 Jun;41(6):2267-2281. doi: 10.1007/s12325-024-02834-9. Epub 2024 Apr 15. PMID 38616241
- [Derived] Mahlangu J, Kaczmarek R, von Drygalski A, Shapiro S, Chou SC, Ozelo MC, Kenet G, Peyvandi F, Wang M, Madan B, Key NS, Laffan M, Dunn AL, Mason J, Quon DV, Symington E, Leavitt AD, Oldenburg J, Chambost H, Reding MT, Jayaram K, Yu H, Mahajan R, Chavele KM, Reddy DB, Henshaw J, Robinson TM, Wong WY, Pipe SW; GENEr8-1 Trial Group. Two-Year Outcomes of Valoctocogene Roxaparvovec Therapy for Hemophilia A. N Engl J Med. 2023 Feb 23;388(8):694-705. doi: 10.1056/NEJMoa2211075. PMID 36812433
- [Derived] Quinn J, Delaney KA, Wong WY, Miesbach W, Bullinger M. Psychometric Validation of the Haemo-QOL-A in Participants with Hemophilia A Treated with Gene Therapy. Patient Relat Outcome Meas. 2022 Jul 18;13:169-180. doi: 10.2147/PROM.S357555. eCollection 2022. PMID 35879931
- [Derived] Ozelo MC, Mahlangu J, Pasi KJ, Giermasz A, Leavitt AD, Laffan M, Symington E, Quon DV, Wang JD, Peerlinck K, Pipe SW, Madan B, Key NS, Pierce GF, O'Mahony B, Kaczmarek R, Henshaw J, Lawal A, Jayaram K, Huang M, Yang X, Wong WY, Kim B; GENEr8-1 Trial Group. Valoctocogene Roxaparvovec Gene Therapy for Hemophilia A. N Engl J Med. 2022 Mar 17;386(11):1013-1025. doi: 10.1056/NEJMoa2113708. PMID 35294811
- [Derived] Rosen S, Tiefenbacher S, Robinson M, Huang M, Srimani J, Mackenzie D, Christianson T, Pasi KJ, Rangarajan S, Symington E, Giermasz A, Pierce GF, Kim B, Zoog SJ, Vettermann C. Activity of transgene-produced B-domain-deleted factor VIII in human plasma following AAV5 gene therapy. Blood. 2020 Nov 26;136(22):2524-2534. doi: 10.1182/blood.2020005683. PMID 32915950

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 48 sites worldwide (United States, Australia, Belgium, Brazil, France, Germany, Israel, Italy, South Korea, South Africa, Spain, Taiwan, and United Kingdom).
Pre-assignment Details: Total of 181 subjects were screened. Of these, 41 subjects were screened without prior participation in 270-902,140 subjects were screened after participating in 270-902. 37 subjects failed screening. Of the remaining 144 enrolled subjects in 270-301,134 were treated with BMN 270. 10 subjects enrolled but were not dosed [5 subjects who did not previously participate in 270-902(direct enrolled population and 5 subjects dosed in 270-301 who previously participated in 270-902(Rollover population)].
Groups:
- BMN 270 (Valoctocogene Roxaparvovec): Single administration of valoctocogene roxaparvovec at a dose of 6E13 vg/kg
  valoctocogene roxaparvovec: Adeno-Associated Virus Vector-Mediated Gene Transfer of Human Factor VIII in Hemophilia A subjects
Period: Overall Study
Arm/Group | BMN 270 (Valoctocogene Roxaparvovec)
Started | 134
Completed (Participants completed Week 104 Visit) | 132
Not Completed | 2
Not completed — Death | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population (n=134): All subjects dosed in 270-301
Arm/Group | BMN 270 (Valoctocogene Roxaparvovec)
Number analyzed (Participants) | 134
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at enrollment, years
  years | 31.7 (10.3)
Age, Customized [Count of Participants; unit: Participants] — Age at enrollment: n(%)
  Participants
    18 to < 30 years | 65
    30 to < 50 years | 56
    >= 50 years | 13
Sex: Female, Male [Count of Participants; unit: Participants] — n(%)
  Percentages were calculated using the total number of subjects (n) in each analysis population as the denominator
  Participants
    Female | 0
    Male | 134
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — n(%)
  Participants
    Hispanic or Latino | 7
    Not Hispanic or Latino | 127
    Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — n(%)
  Participants
    Asian | 19
    Black or African-American | 15
    Native Hawaiian or other Pacific Islander | 1
    White | 96
    Not provided due to patient privacy | 3
Baseline annualized FVIII usage [Mean (Standard Deviation); unit: IU/kg/year] — The annualized utilization (IU/kg/year) of exogenous FVIII replacement therapy is defined as Sum of FVIII use (IU/kg) during calculation period/Total number of days during the calculation period ×365.25.
  IU/kg/year | 4113.69 (1738.92)
Baseline annualized number of FVIII infusions [Mean (Standard Deviation); unit: Infusions/year] — Annualized FVIII infusion rate (count/yr) = (sum(Number of FVIII replacement infusions during calculation period) /sum(follow-up days of the period))*365.25.
  Infusions/year | 137.55 (57.04)
Baseline ABR (all bleeds) [Mean (Standard Deviation); unit: bleeds/year] — All bleeds comprises both treated and non-treated bleeds. In this definition, all bleeds are included, irrespective of treatment with coagulation factors, with the following exception: bleeds due to surgery/procedure are excluded. All bleeds are any reported bleeding events regardless of the use of FVIII or other treatments.
  Annualized bleed rate (episodes/yr) = (sum (number of bleed episodes during calculation period))/(sum (follow-up days of the period)) *365.25
  bleeds/year | 5.97 (11.06)
Baseline ABR (all bleeds) [Count of Participants; unit: Participants] — n(%)
  All bleeds comprises both treated and non-treated bleeds. In this definition, all bleeds are included, irrespective of treatment with coagulation factors, with the following exception: bleeds due to surgery/procedure are excluded. All bleeds are any reported bleeding events regardless of the use of FVIII or other treatments.
  Annualized bleed rate (episodes/yr) = (sum (number of bleed episodes during calculation period))/(sum (follow-up days of the period)) *365.25
  Participants
    0 bleeds/year | 41
    > 0 to 4 | 40
    > 4 to 10 | 31
    > 10 | 22
Baseline ABR (treated bleeds) [Mean (Standard Deviation); unit: bleeds/year] — Bleeds that were treated with FVIII replacement therapy (recorded as "treatment for bleed") within 72 hours and were not associated with surgery or a procedure were included.
  Annualized bleed rate (episodes/yr) = (sum (number of bleed episodes during calculation period))/(sum (follow-up days of the period)) *365.25
  bleeds/year | 5.42 (9.96)
Baseline ABR (treated bleeds) [Count of Participants; unit: Participants] — n(%)
  Bleeds that were treated with FVIII replacement therapy (recorded as "treatment for bleed") within 72 hours and were not associated with surgery or a procedure were included.
  Annualized bleed rate (episodes/yr) = (sum (number of bleed episodes during calculation period))/(sum (follow-up days of the period)) *365.25
  Participants
    0 bleeds/year | 43
    > 0 to 4 | 42
    > 4 to 10 | 29
    > 10 | 20
History of previous diseases [Count of Participants; unit: Participants] — n(%)
  Participants
    Hepatitis B | 20
    Hepatitis C | 41
    HIV | 2
Number of target joints [Count of Participants; unit: Participants] — n(%)
  Target joints are defined as joints with >= 3 spontaneous bleeds (treated or untreated) in the same joint location within any consecutive 6-month (180 days) period in the Baseline period.
  Participants
    0 | 97
    1 | 17
    2 | 9
    3 | 8
    > 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Annualized Number of Bleeding Episodes Irrespective of Exogenous FVIII Replacement Treatment [Annualized Bleeding Rate (ABR) for All Bleeds] in EEP.
Description: All bleeds comprises both treated and non-treated bleeds. In this definition, all bleeds are included, irrespective of treatment with coagulation factors, with the following exception: bleeds due to surgery/procedure are excluded. All bleeds are any reported bleeding events regardless of the use of FVIII or other treatments.
  ABR for all bleeds= Number of bleeding episodes for all bleeds during the calculation period / total number of days during the calculation period * 365.25.
  Baseline: prior to BMN 270 infusion while receiving FVIII prophylaxis.
  EEP: From Week 5 post-BMN 270 infusion (Study Day 33) or the end of FVIII prophylaxis plus the washout period (3 days for products of standard half-life or plasma-derived and 5 days for products of extended half-life), whichever is later, to last visit by the data cut-off for the 2-year analysis, hereafter referred to as "Post FVIII Prophylaxis to Last Visit").
Time Frame: Baseline to efficacy evaluation period (EEP)
Population: Rollover Population (n=112): Subjects who completed approximately 6 months participation in the non-interventional study 270-902 before enrolling in 270-301, were HIV-negative at study screening, and received BMN 270 infusion in 270-301.
Measure: Mean (Standard Deviation); unit: bleeds/year
Arm/Group | BMN 270 (Valoctocogene Roxaparvovec)
Number analyzed (Participants) | 112
bleeds/year | -4.13 (6.93)
Statistical Analysis 1: Comparison: BMN 270 (Valoctocogene Roxaparvovec); Change from baseline in the ABR for all bleeds (post-baseline EEP value - baseline value); Test type: Superiority; p < 0.0001, t-test, 2 sided — P-values were for 2-sided test against 0; Superiority was tested by1-sample t-test to test null hypothesis that change is >=0. Only negative changes represent efficacy; % Reduction from Baseline = -77.0 — 77% reduction

2. Secondary Outcome: Change From Baseline in the Annualized Number of Bleeding Episodes Requiring Exogenous FVIII Replacement Therapy (ABR for Treated Bleeds) in the EEP.
Description: ABR for treated bleeds=Number of bleeding episodes for treated bleeds during the calculation period/total number of days during the calculation period * 365.25
  Bleeds that were treated with FVIII replacement therapy (recorded as "treatment for bleed") within 72 hours and were not associated with surgery or a procedure were included.
  Baseline: prior to BMN 270 infusion while receiving FVIII prophylaxis.
  EEP: From Week 5 post-BMN 270 infusion (Study Day 33) or the end of FVIII prophylaxis plus the washout period (3 days for products of standard half-life or plasma-derived and 5 days for products of extended half-life), whichever is later, to last visit by the data cut-off for the 2-year analysis, hereafter referred to as "Post FVIII Prophylaxis to Last Visit").
Time Frame: Baseline to EEP
Population: Rollover Population
Measure: Mean (Standard Deviation); unit: bleeds/year
Arm/Group | BMN 270 (Valoctocogene Roxaparvovec)
Number analyzed (Participants) | 112
bleeds/year | -4.08 (6.57)

3. Secondary Outcome: Change From Baseline in FVIII Activity at Week 104
Description: The change from baseline (assuming no treatment for severe hemophilia A) in FVIII activity, as measured by chromogenic substrate assay, at Weeks 104 post-BMN 270 infusion.
  Each subject's FVIII activity level at Week 104 is defined as the median of the values obtained at Week 104 with the analysis window defined. The baseline value is imputed as 1 IU/dL for each subject.
  Note: One of the subject's wk104 duplicate data issue was corrected in the 3 year analysis per which the mean (standard deviation) values are reported in outcome measure table.
  Baseline: prior to BMN 270 infusion while receiving FVIII prophylaxis.
Time Frame: Baseline to Week 104
Population: Modified Intent-to-Treat (mITT) Population (n=132): All HIV-negative subjects at study screening who were dosed in 270-301.
Measure: Mean (Standard Deviation); unit: IU/dL
Arm/Group | BMN 270 (Valoctocogene Roxaparvovec)
Number analyzed (Participants) | 132
IU/dL | 21.94 (33.04)

4. Secondary Outcome: Change From Baseline in Annualized FVIII Utilization in EEP.
Description: The change from baseline in the annualized utilization (IU/kg/year) of exogenous FVIII replacement therapy in the Post FVIII Prophylaxis to Last Visit in the EEP.
  The annualized utilization (IU/kg/year) of exogenous FVIII replacement therapy is defined as Sum of FVIII use (IU/kg) during calculation period/Total number of days during the calculation period ×365.25.
  Baseline: prior to BMN 270 infusion while receiving FVIII prophylaxis.
  EEP: From Week 5 post-BMN 270 infusion (Study Day 33) or the end of FVIII prophylaxis plus the washout period (3 days for products of standard half-life or plasma-derived and 5 days for products of extended half-life), whichever is later, to last visit by the data cut-off for the 2-year analysis, hereafter referred to as "Post FVIII Prophylaxis to Last Visit").
Time Frame: Baseline to EEP
Population: Rollover population
Measure: Mean (Standard Deviation); unit: IU/kg/yr
Arm/Group | BMN 270 (Valoctocogene Roxaparvovec)
Number analyzed (Participants) | 112
IU/kg/yr | -3891.27 (1761.16)

5. Secondary Outcome: Change From Baseline in Haemo-QoL-A Quality of Life: Total Score at Week 104
Description: The change from baseline(assuming no treatment for severe hemophilia A) in Haemo-Qol-A score, at wk104 post-BMN 270 infusion.The Haemo-Qol-A questionnaire is a fit for purpose hemophilia-specific health related quality of life(HRQoL)questionnaire for adults consisting of 41 items covering 6 domains(Physical Functioning,Role Functioning,Worry,Consequences of Bleeding,Emotional Impact &Treatment Concerns). The Haemo-Qol-A items are answered on a 6-point Likert scale ranging from 0(none of the time)to 5 (all of the time).The recall period for the Haemo-Qol-A is one month (4-weeks).
  The Haemo-QoL-A domain(physical functioning, role functioning, worry, consequences of bleeding, emotional impact, treatment concern) scores range from 0 to 5 and the total score is derived by summing each domain score (range, 0 to 30). Domain and total scores are transformed to a 0 (minimum) to 100 (maximum) scale with higher scores indicating a better or less impaired haemophilia related quality of life.
Time Frame: Baseline to Week 104
Population: mITT Population: Modified Intent-to-Treat Population - all HIV-negative subjects dosed in 270-301.
  Change from baseline was based on the subjects with available measurements at both time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BMN 270 (Valoctocogene Roxaparvovec)
Number analyzed (Participants) | 126
score on a scale | 7.01 (12.55)

6. Secondary Outcome: Change From Baseline in Haemo-QoL-A Quality of Life: Physical Functioning Domain Score, at Week 104
Description: The change from baseline (assuming no treatment for severe hemophilia A) in Haemo-Qol-A score, at week 104 post-BMN 270 infusion. The Haemo-Qol-A questionnaire is a fit for purpose hemophilia-specific health related quality of life (HRQoL) questionnaire for adults consisting of 41 items covering six domains (Physical Functioning, Role Functioning, Worry, Consequences of Bleeding, Emotional Impact and Treatment Concerns).The Haemo-Qol-A items are answered on a 6-point Likert scale ranging from 0 (none of the time) to 5 (all of the time).The recall period for the Haemo-Qol-A is one month (4-weeks).
  The Haemo-Qol-A physical functioning domain score is an average of each item value within a domain.The range of domain scores is 0 to 5; higher scores mean better HRQoL or less impairment for the domain. The physical functioning domain score is transformed to a 0 (minimum) to 100 (maximum) scale with higher scores indicating a better or less impaired haemophilia-related physical functioning
Time Frame: Baseline to Week 104
Population: mITT population
  Change from baseline was based on the subjects with available measurements at both time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BMN 270 (Valoctocogene Roxaparvovec)
Number analyzed (Participants) | 129
score on a scale | 4.90 (13.78)

7. Secondary Outcome: Change From Baseline in Haemo-QoL-A Quality of Life: Consequences of Bleeding Domain Score, at Week 104
Description: The change from baseline(assuming no treatment for severe hemophilia A)in Haemo-Qol-A score, at week 104 post-BMN 270 infusion. The Haemo-Qol-A questionnaire is a fit for purpose hemophilia-specific health related quality of life(HRQoL)questionnaire for adults consisting of 41 items covering 6 domains(Physical Functioning,Role Functioning,Worry,Consequences of Bleeding,Emotional Impact and Treatment Concerns). The Haemo-Qol-A items are answered on a 6-point Likert scale ranging from 0(none of the time) to 5(all of the time). The recall period for the Haemo-Qol-A is one month (4-wks).
  The Haemo-Qol-A consequences of bleeding domain score is an average of each item value within a domain. The range of domain scores is 0 to 5; higher scores mean better HRQoL or less impairment for the domain. The consequences of bleeding domain score is transformed to a 0 (minimum) to 100 (maximum) scale with higher scores indicating a better or less impaired haemophilia-related consequences of bleeding
Time Frame: Baseline to Week 104
Population: mITT population.
  Change from baseline was based on the subjects with available measurements at both time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BMN 270 (Valoctocogene Roxaparvovec)
Number analyzed (Participants) | 129
score on a scale | 10.29 (17.65)

8. Secondary Outcome: Change From Baseline in Haemo-QoL-A Quality of Life: Role Functioning Domain Score, at Week 104
Description: The change from baseline (assuming no treatment for severe hemophilia A) in Haemo-Qol-A score, at week 104 post-BMN 270 infusion. The Haemo-Qol-A questionnaire is a fit for purpose hemophilia-specific health related quality of life (HRQoL) questionnaire for adults consisting of 41 items covering six domains (Physical Functioning, Role Functioning, Worry, Consequences of Bleeding, Emotional Impact and Treatment Concerns).The Haemo-Qol-A items are answered on a 6-point Likert scale ranging from 0 (none of the time) to 5 (all of the time). The recall period for the Haemo-Qol-A is one month (4-weeks).
  The Haemo-Qol-A role functioning domain score is an average of each item value within a domain. The range of domain scores is 0 to 5; higher scores mean better HRQoL or less impairment for the domain. The role functioning domain score is transformed to a 0 (minimum) to 100 (maximum) scale with higher scores indicating a better or less impaired haemophilia-related role functioning.
Time Frame: Baseline to Week 104
Population: mITT population
  Change from baseline was based on the subjects with available measurements at both time points.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | BMN 270 (Valoctocogene Roxaparvovec)
Number analyzed (Participants) | 128
Score on a scale | 7.37 (15.17)

ADVERSE EVENTS:
Time Frame: Up to data cutoff date 15 November 2021 (Two year data analysis).
Description: Intent-to-Treat (ITT) Population: All subjects dosed in 270-301 study.
Arm/Group | BMN 270 (Valoctocogene Roxaparvovec)
All-Cause Mortality (participants affected / at risk) | 1/134
Serious Adverse Events (participants affected / at risk) | 24/134
Other Adverse Events (participants affected / at risk) | 134/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BMN 270 (Valoctocogene Roxaparvovec) (N=134)
Alanine aminotransferase increased (Investigations) | 2 (2)
Anaphylactic reaction (Immune system disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Gastroenteritis (Infections and infestations) | 2 (2)
Rectal hemorrhage (Gastrointestinal disorders) | 2 (2)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1)
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1)
Cataract (Eye disorders) | 1 (2)
Completed suicide (Psychiatric disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 1 (1)
Hemoperitoneum (Gastrointestinal disorders) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Influenza A virus test positive (Investigations) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Macular hole (Eye disorders) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Peripheral swelling (General disorders) | 1 (1)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pneumonia cytomegaloviral (Infections and infestations) | 1 (1)
Post-procedural hemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Rash maculopapular (Skin and subcutaneous tissue disorders) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (2)
Steroid diabetes (Metabolism and nutrition disorders) | 1 (1)
Traumatic hematoma (Injury, poisoning and procedural complications) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BMN 270 (Valoctocogene Roxaparvovec) (N=134)
Alanine aminotransferase increased (Investigations) | 119 (385)
Aspartate aminotransferase increased (Investigations) | 47 (104)
Weight increased (Investigations) | 22 (36)
Blood creatine phosphokinase increased (Investigations) | 17 (22)
Blood lactate dehydrogenase increased (Investigations) | 9 (14)
Upper respiratory tract infection (Infections and infestations) | 33 (45)
Nasopharyngitis (Infections and infestations) | 29 (52)
Rhinitis (Infections and infestations) | 12 (16)
Folliculitis (Infections and infestations) | 11 (13)
Rash pustular (Infections and infestations) | 11 (12)
Gastroenteritis (Infections and infestations) | 7 (8)
Influenza (Infections and infestations) | 7 (7)
Viral infection (Infections and infestations) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 53 (105)
Back pain (Musculoskeletal and connective tissue disorders) | 25 (32)
Myalgia (Musculoskeletal and connective tissue disorders) | 17 (18)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16 (19)
Arthropathy (Musculoskeletal and connective tissue disorders) | 8 (8)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 (8)
Nausea (Gastrointestinal disorders) | 51 (79)
Diarrhoea (Gastrointestinal disorders) | 28 (43)
Vomiting (Gastrointestinal disorders) | 21 (27)
Dyspepsia (Gastrointestinal disorders) | 11 (13)
Abdominal discomfort (Gastrointestinal disorders) | 10 (10)
Abdominal pain upper (Gastrointestinal disorders) | 10 (15)
Constipation (Gastrointestinal disorders) | 9 (12)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 8 (9)
Fatigue (General disorders) | 40 (53)
Pyrexia (General disorders) | 31 (35)
Pain (General disorders) | 10 (11)
Chills (General disorders) | 9 (9)
Influenza like illness (General disorders) | 7 (8)
Malaise (General disorders) | 7 (8)
Acne (Skin and subcutaneous tissue disorders) | 36 (45)
Rash (Skin and subcutaneous tissue disorders) | 11 (11)
Headache (Nervous system disorders) | 55 (174)
Dizziness (Nervous system disorders) | 9 (14)
Lethargy (Nervous system disorders) | 8 (9)
Migraine (Nervous system disorders) | 7 (8)
Tremor (Nervous system disorders) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 24 (33)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 24 (28)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 9 (10)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Muscle strain (Injury, poisoning and procedural complications) | 13 (19)
Limb injury (Injury, poisoning and procedural complications) | 9 (10)
Contusion (Injury, poisoning and procedural complications) | 8 (11)
Ligament sprain (Injury, poisoning and procedural complications) | 8 (8)
Fall (Injury, poisoning and procedural complications) | 7 (9)
Insomnia (Psychiatric disorders) | 27 (46)
Anxiety (Psychiatric disorders) | 11 (12)
Irritability (Psychiatric disorders) | 7 (8)
Cushingoid (Endocrine disorders) | 16 (16)
Hypertension (Vascular disorders) | 16 (20)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-07-15): https://cdn.clinicaltrials.gov/large-docs/13/NCT03370913/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-13): https://cdn.clinicaltrials.gov/large-docs/13/NCT03370913/SAP_001.pdf